CLINICAL TRIAL: NCT01613690
Title: An Open Label, Non-randomized, Parallel-group Study to Characterize and Compare the Pharmacokinetics, Safety, and Tolerability of a Single Dose of NVA237 in Subjects With Mild, Moderate, Severe and End-stage Renal Impairment With That in Matched Healthy Control Subjects
Brief Title: Comparing the Pharmacokinetics, Safety and Tolerability of NVA237 in Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CNVA237A2105
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-06

CONDITIONS: Renal Impairment
Keywords: Renal impairment; NVA237; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — Glycopyrrolate

ARMS (5):
- Healthy volunteers (Experimental): control group receiving 100 μg NVA237
  Interventions: Drug: NVA237
- Mild renal impairment (Experimental): (eGFR 50-80 mL/min/1.73m2) receiving 100 μg NVA237
  Interventions: Drug: NVA237
- Moderate renal impairment (Experimental): (eGFR 30-49 mL/min/1.73m2) receiving 100 μg NVA237
  Interventions: Drug: NVA237
- Severe renal impairment (Experimental): (eGFR <30 mL/min1.73m2) receiving 100 μg NVA237
  Interventions: Drug: NVA237
- End-stage subjects requiring dialysis (ESRD) (Experimental): receiving 100 μg NVA237
  Interventions: Drug: NVA237

INTERVENTIONS:
Drug: NVA237 — NVA237 is administered via a BREEZHALER device

SUMMARY:
The purpose of this study is to see how the body processes and gets rid of NVA237 in people who have impaired kidney function compared to people whose kidney function is normal.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 to 70 years of age inclusive.
* Female subjects of childbearing potential must be using two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the study, through study completion.
* Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 17 to 35 kg/m2.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent
* For renal insufficient subjects only - Subjects must have stable renal disease without evidence of renal progressive disease (for the purpose of this study stable renal disease will be defined as no significant change for 12 weeks).
* For health subjects only - A serum creatinine within the normal range and an eGFR >80 mL/min/1.73 m2.
* For health subjects only - Matched to at least one renal impaired subjects undergoing study by age (±5 years), sex and weight (±10% BMI).

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months). Smokers will be defined as any subject who reports tobacco use and/or who has a urine cotinine ≥ 500 ng/mL. If non-smoking subject are too difficult to recruit, smokers may be allowed to participate in the study provided they commit to smoke no more than 10 cigarettes/day during the days of PK-assessment
* For healthy subjects, use of any prescription drugs, herbal and fitness/bodybuilding/athletic performance-enhancing supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing
* Recent (within the last three [3] years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting (unless related to water withdrawal during dialysis), palpitations, etc).
* Recent (within the last three [3] years) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* History of multiple and recurring allergies or allergy to the investigational compound/compound class being used in this study.
* Total WBC count which falls outside the range of 3000-12,000/μL, or platelets <100,000/μl at screening.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Concentration of NVA2105 using PK parameter of primary interest - area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter of primary interest - maximum plasma concentration (Cmax) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter of primary interest - renal clearance (CLR) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter of secondary interest - time to Cmax (Tmax) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter of secondary interest - AUC extrapolated to infinity (AUCinf) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter of secondary interest - terminal elimination half-life, determined from plasma concentrations and urinary excretion rates (T1/2) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter of secondary interest - apparent systemic clearance (CL/F) | Day 1, 2, 3, 4 and 5
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Concentration of NVA2105 using PK parameter - amount excreted into the urine from time 0 to 96 h post-dose (Ae0-96h) | Day 1, 2, 3, 4 and 5
  Samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Urine, Analyte: NVA237
Concentration of NVA2105 using PK parameter - T1/2 | Day 1, 2, 3, 4 and 5
  Samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Urine, Analyte: NVA237
Concentration of NVA2105 using PK parameter - CLR | Day 1, 2, 3, 4 and 5
  Samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Urine, Analyte: NVA237

SECONDARY OUTCOMES:
Change in effect of dialysis in End-stage subjects requiring dialysis (ESRD) using PK parameter Cmax | Day 1 of each treatment period
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Change in effect of dialysis in End-stage subjects requiring dialysis using PK parameter AUClast | Day 1 of each treatment period
  Blood samples will be collected at various time points on each visit day; Compound: NVA237 100ug, Matrix: Plasma, Analyte: NVA237
Safety and tolerability of a single inhalation dose of 100μg NVA237 in subjects with mild, moderate, severe, and end-stage renal impairment | Reviewed during each study visit
  Adverse events will be based on evaluation of physical signs, electrocardiograms and clinical laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- See also: Results for CNVA237A2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5583